CLINICAL TRIAL: NCT00820339
Title: Pringle's Maneuver Versus Selective Hepatic Vascular Exclusion in Hepatectomy About Recurrence and Survival :A Prospective Randomized Trial
Brief Title: Pringle's Maneuver Versus Selective Hepatic Vascular Exclusion in Hepatectomy
Acronym: SHVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-002
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; hepatic vein; Surgical resection; occlusion; time to recurrence; overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective Hepatic Vascular Exclusion (Active Comparator): Patients with HCC received Selective Hepatic Vascular Exclusion in hepatectomy.
  Interventions: Procedure: Selective Hepatic Vascular Exclusion
- Pringle's Maneuver (Experimental): Patients with HCC received Pringle's Maneuver in hepatectomy.
  Interventions: Procedure: Pringle's Maneuver

INTERVENTIONS:
Procedure: Selective Hepatic Vascular Exclusion — Inflow occlusion with extraparenchymal control of major hepatic veins results in total liver isolation from the systemic circulation but without interruption of caval flow.
  Other Names: SHVE group
  Arms: Selective Hepatic Vascular Exclusion
Procedure: Pringle's Maneuver — Hepatic pedical clamping is performed by encircling the hepatoduodenal ligament with a tape and then applying a tourniquet or a vascular clamp until the pulse in the hepatic artery disappears distally.
  Other Names: Pringle's Maneuver group
  Arms: Pringle's Maneuver

SUMMARY:
To confirm that SHVE is a safe and effective procedure and it can prevent bleeding of the hepatic vein. To evaluate the recurrence and metastasis in HCC patients undergoing hepatectomy by SHVE.To evaluate that SHVE can improve survival in HCC patients or not.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), a serious disease with high incidence at home and abroad still shows a rising trend. In recent decade, the overall survival rate of the disease has entered a platform stage with little advance despite diversified methods of treatment. The prognosis of HCC is not so satisfying.

Intraoperative bleeding remains a major concern during liver resection. Blood loss usually occurs during parenchymal transection and reperfusion after Pringle's maneuver. The amount of blood loss and the need for blood transfusion have a detrimental effect on the short- and long-term prognosis.

Portal triad clamping is sufficient in most situations to control bleeding during hepatectomy. However, it does not prevent backflow bleeding from hepatic veins, which may become troublesome or even hazardous. This is particularly true in tumors that are large or that have invaded into the branches of the major hepatic veins.

SHVE completely isolates the liver from the systemic circulation with the advantage of preventing backflow hemorrhage or air embolism without having to resort to caval blood flow interruption of THVE.

The purpose of the study is to assess the risk factors for the recurrence and metastasis in HCC patients undergoing hepatectomy by SHVE and to evaluate that SHVE can improve survival in HCC patients or not.

ELIGIBILITY:
Inclusion Criteria:

* Corresponding to diagnostic standards of HCC.
* Patients of liver tumors underwent resection with occlusion of more than one main hepatic veins.
* liver function in the Child-Pugh classification A or B.
* Age between 18~70 years.
* Haven't taken any current treatment.
* Understanding and being willing to sigh the informed consent form.

Exclusion Criteria:

* cannot be follow-up
* severe liver, renal, or brain dysfunction
* with tumor thrombi in the main trunk of portal vein
* with tumor thrombi in the hepatic vein
* with extrahepatic metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1,2,or 3 years

SECONDARY OUTCOMES:
Blood transfusion ,hepatic function of patients after surgery, the incidence rate of complications | 1,2,or 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, M.D., Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China